CLINICAL TRIAL: NCT04993638
Title: Post Market Clinical Follow-up of Dual-mobility Acetabular Cup EUROSCUP MOBILE
Status: Active, not recruiting | Type: Observational
Sponsor: EUROS (Industry)
Responsible Party: Sponsor
Other Study IDs: EC-310-02-01-A
Record Dates: First submitted 2021-06-04; First posted 2021-08-06 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Hip Arthropathy; Hip Osteoarthritis; Hip Arthritis; Hip Fractures; Hip Necrosis; Hip Dysplasia
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Fractures; Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EUROSCUP MOBILE cementless: 107 who received cementless version of EUROSCUP MOBILE
  Interventions: Device: hip arthroplasty
- EUROSCUP MOBILE cemented: 40 who received cemented version of EUROSCUP MOBILE
  Interventions: Device: hip arthroplasty

INTERVENTIONS:
Device: hip arthroplasty — Hip prosthesis surgery

SUMMARY:
EUROSCUP MOBILE is intended for use in primary and revision total hip replacement surgery.

Hip replacement is intended to provide increased patient mobility and reduce pain by replacing the damages hip joint articulation in patients where there is evidence of sufficient sound bone to seat and support the components.

As part of post market vigilance, EUROS will collect data on EUROSCUP MOBILE performances and safety

DETAILED DESCRIPTION:
Post market observational study. This study is retropective and prospective, non comparative.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received EUROSCUP MOBILE.
* Patient informed of its participation to the study
* Patient aged between 18 and 80 years old (<80).

Exclusion Criteria:

* Patient presenting a contraindication to EUROSCUP MOBILE implantation.
* Patient who refused to participate to the study
* Vulnerable subjects

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who fulfill the criteria of eligilibilty according to the instructions for use of EUROSCUP MOBILE
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2034-06-01 (Estimated); Study Completion 2034-06 (Estimated)

PRIMARY OUTCOMES:
Safety of EUROSCUP MOBILE | 1 year
  Collect the safety of the device trought complications occurence rate

SECONDARY OUTCOMES:
Radiological performances of EUROSCUP MOBILE | 1 year
  Collect the performances of the device trought radiological evaluation
Clinical performances of EUROSCUP MOBILE | 1 year
  Collect the performances of the device trought clinical scores
Survival of EUROSCUP MOBILE | 10 year
  Assess the survival rate of the device

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Clinique Montagard, Avignon
  - CHU Gabriel Montpied, Clermont-Ferrand
  - Hôpital Saint Joseph-Saint Luc, Lyon

IPD SHARING:
Plan to Share IPD: No